CLINICAL TRIAL: NCT05792631
Title: A Clinical Study to Compare Caries Detection in Children Between the iTero Element 5D System (NIRI=Near Infra Red Imaging) and Bitewing Radiographs (BWR) as a Diagnostic Aid for the Detection of Primary Carious Lesions Above the Gingiva.
Brief Title: A Study to Compare Caries Detection in the Pediatric Population Between the iTero Element 5D System and Bitewing Radiographs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moti Moskovitz, Prof. Moti Moskovitz DMD, PhD. Director of Postgraduate Program-Dept. of Pediatric Dentistry, Hadassah Medical Center, Faculty of Dental Medicine, Hebrew University of Jerusalem, Israel, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0351-22-HMO
Record Dates: First submitted 2023-01-17; First posted 2023-03-31 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Dental Caries; Patient Compliance
MeSH Terms: conditions — Dental Caries; Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients scheduled for radiographic dental caries assessment (Other): BWR-The most common type of dental x-ray taken during a routine dental checkup is called a "bitewing radiograph." This type of X-ray shows the upper and lower back teeth in a single view and is taken to see how the upper and lower teeth line up, to check for decay, and discover bone loss due to infection and serious gum disease.
  Interventions: Device: Near infra red imaging

INTERVENTIONS:
Device: Near infra red imaging — The iTero Element 5D is an intra-oral scanner that incorporates near-infrared illumination capabilities used to provide a near-infrared image of the teeth enabling the detection of both occlusal and proximal caries, at the various stages, ranging from initial enamel caries to established caries reaching the DEJ.
  Near-infrared Imaging (NIRI) is a nonionizing imaging technology that leverages differences in scattering and absorption of near-infrared light depending on the degree of tooth mineralization.

SUMMARY:
This is a non-significant risk, single site, prospective clinical study. The study will be conducted in the department of pediatric dentistry of the faculty of dental medicine of the Hebrew university, Israel

DETAILED DESCRIPTION:
This is a non-significant risk, single site, prospective study to be conducted in the department of pediatric dentistry of the Hadassah Medical Center, Faculty of Dental Medicine, Hebrew University of Jerusalem, Israel. Subject participation will require one visit during which consent, screening, enrollment, and imaging will be performed.

Clinical and diagnostic methods to be used during this study are those that are routinely used in the diagnosis of caries in this site, which include bitewing radiographs (BWR). This standard of care is provided for all site's patients, including the patients who don't participate in this clinical study.

A standard set of BWR for subjects ages 4-9 years will be taken to include the complete dentition of the subjects. No additional x-ray should be taken for the sole purpose of this trial.

In addition to the routine clinical diagnostics, the subjects will be scanned using the 5D system. The investigator will capture a full arch scan of the maxillary arch and mandibular arch of each subject with the iTero Element 5D system. For each subject, the Investigator will grade carious lesions in the BWR and Element intra-oral scan according to ADA staging guidelines. The results will be documented using Caries Evaluation Forms. The Investigator will assess and document the findings of each diagnostic test separately before reviewing the next test.

In cases where caries debridement is indicated, carious lesion depth will be documented during and compared to NIRI and BWR images.

All treatment decisions will be made according to the standard of care in the clinic and no treatment will be conducted for the sole purpose of the study

ELIGIBILITY:
Inclusion Criteria:

* Ages 4-9 years
* Subjects scheduled for bilateral BWR as part of their standard of care
* Subjects with a recent bilateral BWR which were obtained up to 14 days prior to study visit

Exclusion Criteria:

* Subjects who have been diagnosed with epilepsy
* Subjects with a known allergy to latex or plastic
* Subjects with allergies to any dental or oral health products
* Subjects who have undergone a dental treatment since the acquisition of the recent bilateral BWR

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the iTero 5D compared to BWR in dental caries detection | Grading the carious lesions for the first 20 subjects will be conducted up to 2 month from completion the first 20 subjects visits. The rest 50 subjects will be evaluated up to 1 month from completion the last subject visit.
  For each subject, the Investigator will grade carious lesions in the BWR and Element intra-oral scan (NIRI) according to ADA staging guidelines. The results will be documented using Caries Evaluation Forms for BWR and for Element intra-oral scan . The Investigator will assess and document the findings of each diagnostic test separately before reviewing the next test.
  The iTero 5D performance will be non-inferior to BWR performance in detecting the existence of primary interproximal caries lesions above the gingiva in pediatric population.
  The study will include an interim analysis to assess the iTero Element 5D system usability among the first 20 pediatric subjects.

SECONDARY OUTCOMES:
To compare users' experience using a qualitative questionnaire | The questionnaire will be filled immediately after the intra-oral scan for each subject. Final report of the comparison will be generated up to 15 weeks from last subject visit.
  Qualitative users' feedback will be collected through questionnaire relating to: chair time, the ability to capture tooth surfaces (reachability), patient's experience (gag reflex, discomfort),what Frankl rating would reflect the patient's behavior during the procedure,what is the patient legal guardian's compliance to approve the procedure, if and how the 3D model of the scan assists as a patient communication tool

OTHER OUTCOMES:
To compare carious lesions depth as appears in NIRI and BWR images to clinical depth observed during caries excavation | During the study period and up to 6 months from last subject visit
  Lesion depth will be documented in cases where caries debridement was conducted. NIRI and BWR images will be compared to the clinical findings

CONTACTS AND LOCATIONS:
Overall Officials: Moti Moskovitz, Prof., Principal Investigator — Hadassah Medical Center, Faculty of Dental Medicine, Hebrew University of Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT05792631/Prot_SAP_000.pdf